CLINICAL TRIAL: NCT03727919
Title: A Temporal Analysis of the Robustness of Hemiplegic Gait and Standing Balance Early After sTroke - the TARGET Research Project
Brief Title: Exoskeleton-assisted Training to Accelerate Walking Recovery Early After Stroke: the TARGET Phase II Study
Acronym: TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Jonas Schröder, Principle investigator, PhD researcher, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-2; 1S64819N (Other Grant/Funding Number: Fonds Wetenschappelijk Onderzoek (Brussel, Flanders))
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Stroke; Paresis; Gait, Hemiplegic
Keywords: stroke; rehabilitation; robotics
MeSH Terms: conditions — Stroke; Paresis; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the "early group" or "delayed group". Both groups will be provided a dose- and content-controlled intervention in addition to usual care. The early group will receive this intervention at approximately 2 weeks post-stroke and the delayed group at 8 weeks post-stroke. As such, this study is explicitly designed to investigate the effects of time to initiate rehabilitation on recovery outcomes.
Who Masked: Outcomes Assessor
Masking Description: A blinded assessor will be allocated to a certain participant when she/he was succesfully enrolled. This means that the same assessor will perform the clinical assessments (i.e., FAC, 10-m Walk Test, FM, MI) at the different measurement occasions for this participant to avoid inter-assessor variability effects on longitudinal recovery trajectories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Experimental Group (Experimental): N = 20 Intervention = 1-hour sessions of exoskeleton-assisted gait training, using the Ekso GT (Ekso Bionics, CA, USA) in addition to standard care Frequency = 4 times per week for 4 weeks, provided within the first 6 weeks post-stroke
  Interventions: Behavioral: Exoskeleton-assisted gait training
- Delayed Experimental Group (Experimental): N = 20 Intervention = 1-hour sessions of exoskeleton-assisted gait training, using the Ekso GT (Ekso Bionics, CA, USA) in addition to standard care Frequency = 4 times per week for 4 weeks, provided between week 8 and week 12 post-stroke
  Interventions: Behavioral: Exoskeleton-assisted gait training

INTERVENTIONS:
Behavioral: Exoskeleton-assisted gait training — In the experimental groups, participants are provided with 1-hour sessions of gait training with robot assistance, 4 times per week for 4 weeks. Assistance is provided by the Ekso GT (Ekso Bionics, Richmond, CA, USA), an exoskeleton consisting of fitted metal braces that supports the legs, feet, and trunk of the patient. Powered motors drive knee and hip joints in the sagittal plane to assist during standing up and walking over level surfaces. Steps are initiated if an active weight-shift towards the stance leg is performed by the patient. The provided assistance in stance and swing is adaptable to the patient's ability and can be adjusted for each leg separately.

SUMMARY:
Phase II: Investigating the effects of additional robot-assisted gait training either initiated early (2 weeks post-stroke) or delayed (8 weeks post-stroke) after stroke onset.

DETAILED DESCRIPTION:
GENERAL:

Pre-clinical research has pointed towards a time window of enhanced responsiveness to therapy early after stroke. For example, training has led to substantial recovery if initiated 5 or 14, but not 30 days post-stroke in a rodent model (Biernaski 2004). It is suggested that this early period is characterized by heightened levels of plasticity and that training can exploit this leading to improved outcome. The typically observed non-linear recovery pattern in stroke survivors (Kwakkel 2004) might suggest that similar mechanisms are induced in the human brain, however clinical research on this is disappointingly sparse.

In two closely inter-related phases, we aim to examine the biomechanical changes related to walking recovery in general (Phase I) and the specific effects of robot-assisted training (Phase II). By that, we aim to detect a time window in stroke survivors which resembles the same characteristics as observed in animal models. To initiate gait training at an early stage, when patients usually present severe weakness and balance deficits, a mobile exoskeleton is used which is developed to provide intensive walking practice.

OBJECTIVES:

(II.a) Are stroke survivors who train with the assistance of a robot at an early stage more likely to achieve independent walking?

(II.b) Does additional robot-assisted training modulate the recovery of standing and walking ability by enhancing behavioral restitution?

ELIGIBILITY:
Inclusion Criteria:

* First-ever, MRI- or CT-confirmed, ischemic or hemorrhagic, anterior circulation stroke
* Age: 18 - 90 years
* Baseline assessments within the first 14 days after stroke onset
* Unable to walk independently at baseline (FAC <3)
* Moderate to severe weakness of the lower limb at baseline (MI </=75)
* Pre-morbid independence in activities of daily living (mRS </=2) and gait (FAC >3)
* Able to communicate and comprehend
* Sufficient motivation to participate
* Provided a written informed consent

Exclusion Criteria:

* No other neurological condition affecting motor functions of the lower limbs
* Pre-existing musculoskeletal impairment severely affecting the gait pattern
* Body weight > 100 kg
* Severe spasticity or contractures that prevent safe use of the exoskeleton
* Medically unstable to participate in additional therapy sessions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Change on the Fugl Meyer motor assessment - subscale lower extremity (FM-LE) | Longitudinal change is determined between the following time points: Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  This scale measures the level of of volitional, selective control of muscles of the paretic lower limb.
  Scoring: This scale is scored from 0 (no reflex activity) to 34 (volitional movement out of synergies).

SECONDARY OUTCOMES:
Trunk Control Test - item sitting balance | Baseline (0-1 week post-stroke)
  Sitting balance is part of the prognostic model used to stratify patients at baseline.
  Scoring: 0 - 1 (able to sit independently without support of the legs or trunk 30 seconds)
Motricity Index - subscale lower extremity (MI-LE) | Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  Strength of major muscle groups of the paretic lower limb is assessed. At baseline this is part of the prognostic model used to stratify patients.
  Scoring: This scale is scored from 0 (no muscle activity) to 99 (normal strength over full range of motion in hip flexors, knee extensors and ankle dorsiflexors).
Berg Balance Scale - item standing unsupported | Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  This item of the BBS indicates the ability to stand independently and therefore reflects the process of functional walking recovery within the first 6 months post-stroke.
  Scoring: This scale includes 5 levels (0-4), ranging from "unable to stand 30 seconds unassisted" (0) to "able to stand safely 2 minutes" (5).
Functional Ambulation Categories (FAC) | Baseline (0-1 week post-stroke), 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  This scale indicates the ability to walk independently and therefore reflects the process of functional walking recovery within the first 6 months post-stroke.
  Scoring: This scale includes 6 levels (0-5), ranging from "nonfunctional ambulation" (0) to "ambulate independently, on level and non-level surfaces including stairs and inclines" (5).
Kinetic analyses of standing balance & gait | 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  Dual-force plate measurements are able to indicate the adopted control strategies for standing balance and walking. These analyses are used to distinguish between behavioral restitution and the use of compensation strategies.
EMG analyses of standing balance & gait | 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke
  EMG analyses will be performed to gain insights in the muscle recruitment of patients during standing and walking. These analyses are used to distinguish between behavioral restitution and the use of compensation strategies.
Spatio-temporal analyses of gait | 3 weeks post-stroke, 5 weeks post-stroke, 8 weeks post-stroke, 12 weeks post-stroke, 24 weeks post-stroke.
  Assessing comfortable (self-selected) speed and spatial/temporal symmetry of gait over a short distance.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Schröder, PhD Student, Principal Investigator — Dept. Rehabilitation Sciences & Physiotherapy, University of Antwerp, Belgium; Wim Saeys, Prof. Dr., Study Chair — Dept. Rehabilitation Sciences & Physiotherapy, University of Antwerp, Belgium; Steven Truijen, Prof. Dr., Study Director — Dept. Rehabilitation Sciences & Physiotherapy, University of Antwerp, Belgium
Locations (3):
- Belgium (3):
  - GZA Ziekenhuis - campus St Augustinus & Campus St Vincentius, Wilrijk, Antwerp
  - Antwerp University Hospital, Antwerp
  - RevArte Rehabilitation Hospital, Antwerp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroder J, Yperzeele L, Embrechts E, Loureiro-Chaves R, Hallemans A, Lafosse C, Truijen S, Kwakkel G, Saeys W. Exoskeleton-assisted training to enhance lower limb motor recovery in subacute stroke: does timing matter? A pilot randomized trial. Front Stroke. 2024 May 14;3:1379083. doi: 10.3389/fstro.2024.1379083. eCollection 2024. PMID 41542275